CLINICAL TRIAL: NCT06675123
Title: A Pilot Study of Pacritinib Combined With a BTK Inhibitor in Patients With Relapsed/Refractory Mantle Cell Lymphoma
Brief Title: Pacritinib in Combination With a BTK Inhibitor for the Treatment of Patients With Relapsed or Refractory Mantle Cell Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23184; NCI-2024-08854 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23184 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Mantle Cell Lymphoma; Refractory Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Biopsy; Specimen Handling; 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pacritinib, BTK inhibitor) (Experimental): Patients receive pacritinib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also continue to receive BTK inhibitor per standard of care. Additionally, patients undergo blood sample collection, optional tissue biopsy, bone marrow biopsy and aspiration and PET/CT throughout the study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: BTK Inhibitor; Procedure: Computed Tomography; Drug: Pacritinib; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biopsy — Undergo optional tissue biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow biopsy and aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and aspiration
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: BTK Inhibitor — Given BTK inhibitor
  Other Names: Tyrosine-Protein Kinase BTK Protein
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Pacritinib — Given PO
  Other Names: Oral JAK2 Inhibitor SB1518; SB 1518; SB-1518; SB1518
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase I trial tests the safety and side effects of pacritinib in combination with a Bruton's tyrosine kinase (BTK) inhibitor and how well it works in treating patients with mantle cell lymphoma that has come back after a period of improvement (relapsed) or that has not responded to previous treatment (refractory). Pacritinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. BTK inhibitors block a protein called BTK which is present on B-cell (a type of white blood cell) cancers such as mantle cell lymphoma at abnormal levels. This may help keep tumor cells from growing and spreading. Giving pacritinib in combination with a BTK inhibitor may be safe, tolerable and/or effective in treating patients with relapsed or refractory mantle cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Obtain a preliminary estimate of the safety and tolerability of the combination of pacritinib with a covalent BTK inhibitor (e.g., ibrutinib, acalabrutinib, zanubrutinib) in patients with relapsed/refractory (R/R) mantle cell lymphoma (MCL).

SECONDARY OBJECTIVES:

I. Obtain a preliminary estimate of the overall response rate (ORR) of the combination of pacritinib with a BTK inhibitor in patients with R/R MCL.

II. Obtain a preliminary estimate of the duration of response and progression-free survival in patients with R/R MCL treated with a combination of pacritinib with a BTK inhibitor.

EXPLORATORY OBJECTIVES:

I. Explore the association between clinical outcomes, elimination of tumor associated macrophages (TAMs), and expression of IL-10.

II. Evaluate minimal residual disease (MRD) in patients who obtain a complete metabolic response to therapy.

OUTLINE:

Patients receive pacritinib orally (PO) twice daily (BID) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also continue to receive BTK inhibitor per standard of care. Additionally, patients undergo blood sample collection, optional tissue biopsy, bone marrow biopsy and aspiration and positron emission tomography (PET)/computed tomography (CT) throughout the study.

After completion of study treatment, patients are followed up at 30 days. Patients without progression are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Be willing to provide tissue from a fresh core or excisional biopsy (performed as standard of care) of a tumor lesion prior to starting study therapy or from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Age: ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Histologically confirmed diagnosis of mantle cell lymphoma according to the World Health Organization (WHO) classification with a characteristic immunophenotypic profile with CD5+, CD20+, and with either cyclin D1 expression by immunohistochemistry (IHC), or positive by fluorescence in situ hybridization (FISH) or cytogenetics for the t(11,14) translocation, or both. Patients whose tumor is negative for cyclin D1 expression are allowed providing hemato-pathology confirmation of the diagnosis of MCL

  * Relapsed or refractory disease after at least 1 prior line of systemic therapy
  * Relapse must have been confirmed histologically with hematopathology review. Exceptions may be granted with study PI approval
* Patient must be receiving treatment with single agent ibrutinib or another covalent BTK inhibitor (e.g., acalabrutinib, zanubrutinib), and must have previously achieved complete response (CR) or partial response (PR) to the BTK inhibitor, and must show evidence of progressive MCL at the time of enrollment
* Radiographically measurable disease by Lugano criteria (e.g., one or more nodal sites of disease ≥ 1.5 cm and/or extranodal sites of disease ≥ 1.0 cm in longest dimension)

  * If measurable bone marrow involvement or circulating disease has been confirmed in the absence of radiographically measurable disease, exceptions may be granted with study PI approval
* Fully recovered from the acute toxic effects (except alopecia) to ≤ grade 1 to prior anti-cancer therapy
* WITHOUT BONE MARROW INVOLVEMENT: Absolute neutrophil count (ANC) ≥ 1,000/mm^3

  * NOTE: Growth factor is not permitted within 7 days of ANC assessment unless cytopenia is secondary to disease involvement
* WITH BONE MARROW INVOLVEMENT: ANC ≥ 500/mm^3

  * NOTE: Growth factor is not permitted within 7 days of ANC assessment unless cytopenia is secondary to disease involvement
* WITHOUT BONE MARROW INVOLVEMENT: Platelets ≥ 75,000/mm^3

  * NOTE: Platelet transfusions are not permitted within 7 days of platelet assessment unless cytopenia is secondary to disease involvement
* WITH BONE MARROW INVOLVEMENT: Platelets ≥ 25,000/mm^3

  * NOTE: Platelet transfusions are not permitted within 7 days of platelet assessment unless cytopenia is secondary to disease involvement
* Total bilirubin ≤ 4 x upper limit of normal (ULN) (If hepatic involvement by lymphoma, or Gilbert's disease: ≤ 3 x ULN)
* Aspartate aminotransferase (AST) ≤ 3 x ULN (If hepatic involvement by lymphoma: AST ≤ 5 x ULN)
* Alanine aminotransferase (ALT) ≤ 3 x ULN (If hepatic involvement by lymphoma: ALT ≤ 5 x ULN)
* Creatinine clearance of ≥ 30 mL/min per 24 hour urine test or the Cockcroft-Gault formula
* IF NOT RECEIVING ANTICOAGULANTS: International normalized ratio (INR) OR prothrombin (PT) ≤ 1.5 x ULN
* IF ON ANTICOAGULANT THERAPY: PT must be within therapeutic range of intended use of anticoagulants
* IF NOT RECEIVING ANTICOAGULANTS: Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN
* Left ventricular ejection fraction (LVEF) ≥ 50%
* Mean corrected QT interval (QTc) (calculated from 3 electrocardiograms using Fridericia formula) ≤ 480 ms
* WOMEN OF CHILDBEARING POTENTIAL: (WOCBP): Negative urine or serum pregnancy test

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to abstain from heterosexual intercourse or use a highly effective method of birth control (defined as those resulting in a failure rate of < 1% per year) during the treatment period until at least 90 days after the last dose of pacritinib and until at least 30 days after the last dose of BTK inhibitor

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only) with no identified cause other than menopause
  * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormone releasing intrauterine devices, and copper intrauterine devices. Note that oral contraceptives or progestin injection (e.g., Depo-Provera) alone are not considered highly effective methods of contraception on their own in combination with pacritinib; an additional barrier method (diaphragm with spermicidal gel or condoms with spermicide), double-barrier methods (diaphragm with spermicidal gel and condoms with spermicide), partner vasectomy, or total abstinence are required

Exclusion Criteria:

* Autologous hematopoietic stem cell transplant within 3 months of day 1 of protocol therapy
* Prior allogeneic stem cell transplant
* Prior treatment with pacritinib or a janus kinase 2 (JAK2) inhibitor
* Concomitant treatment with pirtobrutinib
* Strong CYP3A4 inducers/ inhibitors within 14 days prior to day 1 of protocol therapy

  * Note: Shorter washout periods may be permitted with approval of the study PI, provided that the washout period is at least five half-lives of the drug prior to day 1 of protocol therapy
* Systemic treatment with medications that increase the risk of bleeding, including anticoagulants, antiplatelet agents (except for aspirin dosages of ≤ 100 mg per day), anti-vascular endothelial growth factor (anti-VEGF) agents, and daily use of cytochrome C oxidase subunit 1 (COX-1) inhibiting non-steroidal anti-inflammatory drugs (NSAIDs) within 14 days prior to day 1 of protocol therapy
* Systemic treatment with medications with arrhythmogenic potential within 14 days prior to day 1 of protocol therapy. Shorter washout periods may be permitted with approval of the study PI, provided that the washout period is at least five half-lives of the drug prior to day 1 of protocol therapy
* Systemic steroid therapy for any cause must be tapered down to ≤ 20 mg/day prednisone or equivalent. Exceptions are:

  * Use of brief (≤ 7 days) course of high dose corticosteroids (100 mg/day prednisone or equivalent) prior to initiation of study therapy for control of lymphoma-related symptoms
  * Inhaled or topical steroids
  * Use of mineralocorticoids for management of orthostatic hypotension
  * Use of physiologic doses of corticosteroids for management of adrenal insufficiency
* Significant recent bleeding history defined as National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade ≥ 2 within 3 months prior to day 1 of protocol therapy, unless precipitated by an inciting event (e.g., surgery, trauma, or injury)
* Known bleeding disorders (e.g., von Willebrand's disease or hemophilia)
* Factors that increase the risk for QT interval prolongation (eg, hypokalemia [defined as serum potassium < 3.0 mEq/L that is persistent and refractory to correction], or history of long QT interval syndrome)
* Clinically significant cardiovascular disease such as symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 3 months of screening, any class III or IV cardiac disease as defined by the New York Heart Association (NYHA) Functional Classification, or any class C or D cardiac disease as defined by the NYHA Objective Assessment

  * Note: Subjects with controlled, asymptomatic atrial fibrillation/flutter can enroll on study
* Inability to swallow and retain an oral medication
* Any active gastro-intestinal or metabolic condition that could significantly interfere with absorption of oral medication
* Active or uncontrolled inflammatory or chronic functional bowel disorder such as Crohn's disease, inflammatory bowel disease, chronic diarrhea, or chronic constipation
* Known hypersensitivity to compounds of similar chemical composition to study agent or any of the following inactive ingredients: microcrystalline cellulose, polyethylene glycol, and magnesium stearate, or to loperamide or equivalent antidiarrheal medication
* Known active central nervous system (CNS) involvement by lymphoma, including leptomeningeal involvement
* Known history of progressive multifocal leukoencephalopathy (PML)
* Prior or concurrent malignancy whose natural history or treatment could interfere with the safety or efficacy assessment of the protocol therapy
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment or any major episode of infection (as evaluated by the investigator) within 4 weeks prior to day 1 of protocol therapy
* Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. Testing to be done only in patients suspected of having infections or exposures. Patients with history of HBV infection (defined as negative hepatitis B surface antigen [HBsAg] and positive hepatitis B core antibody [HBcAb]) are eligible if HBV deoxyribonucleic acid (DNA) is undetectable, if they are willing to undergo DNA testing on day 1 of every cycle and every three months for at least 12 months after the last cycle of study treatment and appropriate antiviral therapy. Patients who are positive for HCV antibody are eligible if polymerase chain reaction (PCR) is negative for HCV RNA (PCR testing only required if HCV antibody testing is positive).
* Known active human immunodeficiency virus (HIV) infection. Subjects who have an undetectable or unquantifiable HIV viral load with CD4 > 200 and are on highly active antiretroviral therapy (HAART) medication are allowed. Testing to be done only in patients suspected of having infections or exposures
* FEMALES ONLY: Pregnant or breastfeeding
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-03-08 (Estimated); Study Completion 2028-03-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days after last dose of study drug
  Will be graded using National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. AEs will be summarized by type, severity, and attribution.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up 12 months
  Will be defined as the proportion of response evaluable participants that achieve a best response of either complete metabolic response (CMR) or partial metabolic response (PMR) after the start of protocol therapy and prior to disease progression and/or start of other anti-lymphoma therapy. ORR will be estimated along with the 95% exact binomial confidence interval.
Duration of response (DOR) | From the first achievement of PMR or CMR to time of progressive disease or death, whichever is earlier, assessed up to 12 months
  DOR will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error, 95% confidence interval will be constructed based on log-log transformation. Median DOR will be estimated when available. Descriptive analyses may be done separately for particular Bruton's tyrosine kinase (BTK) inhibitor(s) depending on the number of patients treated.
Progression-free survival (PFS) | From start of protocol treatment to time of disease relapse/progression or death due to any cause, whichever occurs earlier, assessed up to 12 months
  PFS will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error, 95% confidence interval will be constructed based on log-log transformation. Median PFS will be estimated when available. Descriptive analyses may be done separately for particular BTK inhibitor(s) depending on the number of patients treated.

CONTACTS AND LOCATIONS:
Overall Officials: Tycel J Phillips, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States